CLINICAL TRIAL: NCT01313026
Title: Treatment of "Low Anterior Resection Syndrome" by Percutaneous Nerve Evaluation and Transanal Irrigation. A Randomized Cross Over Study.
Brief Title: Treatment of "Low Anterior Resection Syndrome" by Percutaneous Nerve Evaluation and Transanal Irrigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to recruit participants
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LARS 001
Record Dates: First submitted 2011-01-07; First posted 2011-03-11 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-06

CONDITIONS: Rectal Cancer
Keywords: Percutaneous nerve evaluation; Transanal irrigation; Low anterior resection syndrome
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PNE first (Active Comparator): patients randomised to start with PNE stimulation over 4 weeks. Then the stimulator will be removed and after a wash out period of 4 weeks they will be trained in transanal irrigation
  Interventions: Procedure: Percutaneous nerve evaluation
- TAI first (Active Comparator): Patients randomised to start with transanal irrigation treatment in 8 weeks, thereafter a wash out period of 4 weeks before being implanted with a neuro stimulator
  Interventions: Procedure: Percutaneous nerve evaluation

INTERVENTIONS:
Procedure: Percutaneous nerve evaluation — Implantation of a nerve stimulator to stimulate the sacral nerve plexus
  Other Names: The Peristeen Anal Irrigation System; Medtronic nerve stimulators

SUMMARY:
A randomised trial testing the effect of percutaneous nerve evaluation and transanal irrigation on bowel function in patients after low anterior resection for rectal cancer.

DETAILED DESCRIPTION:
Patients will undergo anal physiological assessment and will then be randomized to either treatment arm. The first 12 weeks they will be optimized in the conservative treatment of their bowel function before beginning active treatment with TAI or PNE. After 8 and 4 weeks respectively, the treatment will stop and they will have a period of 4 weeks back on optimized conservative treatment before beginning active treatment in the other active arm.

Detailed records of bowel, micturition and sexual function and QoL will be obtained at regular intervals during the entire trial fase.

ELIGIBILITY:
Inclusion Criteria:

* Low anterior resection for rectal cancer between May 2001 and May 2011

Exclusion Criteria:

* Non-radical resection
* metastatic disease
* Chemotherapy
* Radiotherapy
* Previously treated for another cancer
* Dementia or other mental retardation/severe mental disease
* Inability to read and understand the Danish language
* Recurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2018-02 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
changes in LARS score | baseline, 12, 16, 20, 24 and 28 weeks
  A symptom score ranging from 0 to 42 points calculated on the basis of bowel function

SECONDARY OUTCOMES:
Sexual function | baseline, 12, 16, 20, 24 and 28 weeks
  self-reported sexual function measured by validated questionnaires
Bladder function | baseline, 12, 16, 20, 24 and 28 weeks
  self-reported bladder function by validated questionnaires
Incontinence | baseline, 12, 16, 20, 24 and 28 weeks
  faecal incontinence measured by wexner score and St. Marks incontinence score
Patient Satisfaction | baseline, 12, 16, 20, 24 and 28 weeks
  patient satisfaction measured on a VAS

CONTACTS AND LOCATIONS:
Overall Officials: Katrine J. Emmertsen, MD, Principal Investigator — University of Aarhus
Locations (1):
- Colorectal Surgical Department P, Aarhus University Hospital, Aarhus, Denmark